CLINICAL TRIAL: NCT04691687
Title: OUTpatient Intravenous LASix Trial in Reducing Hospitalization for ADHF (OUTLAST)
Brief Title: OUTpatient Intravenous LASix Trial in Reducing Hospitalization for Acute Decompensated Heart Failure
Acronym: OUTLAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Dr John Heitner, Co-Director of Cardiovascular Research, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 307139; 307139 (Other: New York-Presbyterian Brooklyn Methodist Hospital)
Record Dates: First submitted 2020-12-23; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
Keywords: heart failure; hospitalization; diuretics; IV diuretics; mortality
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: A single center prospective randomized double-blind controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects, nurses and treating physicians will be blinded to whether the subjects are receiving continuous IV furosemide (group 2) or continuous IV placebo (group 3). The pharmacist will not be blinded to help administer the appropriate medication. Because the trial will be double-blinded, safety laboratory tests will be performed for each subject for the duration of the trial, regardless of the treatment arm, and will be monitored by the research coordinator. Similarly, monitoring of potential side effects will be continuous and irrespective of treatment assignment. Outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (Group 1) (No Intervention): Patients in Group 1 received standard of care treatment per heart failure guidelines at the discretion of the primary cardiologist involved in the patient's care.
- IV Placebo Infusion (Placebo Comparator): Patients in Group 2 received IV saline infusion (20-40 ml) concentrated by the pharmacist to minimize fluid intake.The infusions were continuous over 3 hours, biweekly over a one-month period.
  Interventions: Drug: IV Solution
- IV Furosemide Infusion (Experimental): The dose assignments were categorized into low dose (20 mg bolus with 20 mg/hour infusion sessions and 2 ml saline), intermediate dose (40 mg bolus with 40 mg/hour infusion sessions and 4 ml saline) and high dose (80 mg bolus with 80 mg/hour infusion sessions). The infusions were continuous over 3 hours, biweekly over a one-month period.Infusions were held at the discretion of the physician utilizing a written protocol (creatinine 25% above baseline, SBP <80 mmHg or symptoms of presyncope).
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — IV loop diuretic therapy
  Other Names: IV Furosemide
  Arms: IV Furosemide Infusion
Drug: IV Solution — IV Placebo comparator
  Other Names: IV Normal Saline 0.9%
  Arms: IV Placebo Infusion

SUMMARY:
Single-center, prospective double-blinded randomized control trial to evaluate the the feasibility, efficacy and safety of outpatient IV diuretic therapy in treatment of heart failure.

DETAILED DESCRIPTION:
Patients were randomized by a clinical pharmacist with the ratio of 1:1:1 into 3 groups: standard of care control arm (Group 1), IV placebo infusion (Group 2), and IV furosemide infusion (Group 3).Patients in Group 2 and 3 received a comprehensive Heart Failure (HF)-care protocol that included bi-weekly clinic visits for dose-adjusted IV-diuretics, medication adjustment and education. Patients, nurses and treating physicians were blinded to the randomization. Patients in Group 1 received standard of care treatment per heart failure guidelines at the discretion of the primary cardiologist involved in the patient's care.8 Patients in Group 2 received IV saline infusion (20-40 ml) concentrated by the pharmacist to minimize fluid intake. Patients in Group 3 received IV furosemide calculated by the pharmacist to be equivalent or higher in dose compared to the patient's home oral dose. The dose assignments were categorized into low dose (20 mg bolus with 20 mg/hour infusion sessions and 2 ml saline), intermediate dose (40 mg bolus with 40 mg/hour infusion sessions and 4 ml saline) and high dose (80 mg bolus with 80 mg/hour infusion sessions). The infusions were continuous over 3 hours, biweekly over a one-month period. Infusions were held at the discretion of the physician utilizing a written protocol (creatinine 25% above baseline, Systolic Blood Pressure(SBP) <80 mmHg or symptoms of presyncope). Patients in both Groups 2 and 3 resumed all of their oral home medications for HF post infusion visits per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients being admitted with ADHF over 18 years old
* Known history of systolic or diastolic dysfunction of greater than 6 weeks
* NYHA Class II-IV
* Heart failure as defined in [Table 1]. One symptom must be present at time of screening and one sign must be present in the last 12 months
* Elevated pro-BNP >/= 360 pg/ml and not explained by any other etiology
* Willing to consent and comply with scheduled visits and phone calls

Table 1. Criteria for Diagnosing Heart Failure

SYMPTOMS (at least 1 must be present at time of screening):

* Paroxysmal nocturnal dyspnea
* Orthopnea
* Dyspnea on mild or moderate exertion

SIGNS (at least 1 must be present in the last 12 months)

* Any rales post cough
* Jugular venous pressure >/= 10 cm H20
* Lower extremity edema
* Chest X-Ray (CXR) demonstrating pleural effusion, pulmonary congestion, or cardiomegaly

Exclusion Criteria:

* Systolic blood pressure <85 mmHg
* Signs of significant respiratory distress, according to the discretion of the investigator.
* Biventricular Implantable Cardioverter-Defibrillator(ICD) placement within 15 days, cardiogenic shock or volume depletion
* Chronic dialysis
* Acute renal failure defined as creatinine > 2 x baseline
* Severe systemic illness with life expectancy judged less than three years
* Chronic pulmonary disease requiring home O2, oral steroid therapy or hospitalization for exacerbation within 12 months, or significant chronic pulmonary disease in the opinion of the investigator
* Primary hemodynamically significant uncorrected valvular heart disease, obstructive, or regurgitant, or any valvular disease expected to lead to surgery during the trial.
* Atrial fibrillation with resting heart rate >90 bpm
* Myocardial infarction in past 90 days
* Percutaneous coronary intervention in past 30 days
* Heart transplant recipient or currently implanted left ventricular assist device
* Stroke in past 90 days
* No acute infection especially requiring IV antibiotics
* Allergy to Lasix
* Known chronic hepatic disease, defined as aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels > 3.0 times the upper limit of normal
* Non-verbal patients, patients who cannot speak or understand English, patients with dementia and psychiatric illness, patients who are blind or deaf and patients who are transferred to different hospital will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Re-hospitalization for Heart Failure | 30 days
  30-day rehospitalization for Heart Failure

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire(KCCQ) outcome measures | Change from Baseline to 30 days
  Change in Quality of life will be quantified using KCCQ questionnaires
Death, Myocardial Infarction, Stroke | 30 days, 180 days
  Occurrence of death, myocardial infarction, or stroke
PHQ-2 outcome measures | Change from Baseline to 30 days
  Change in depressive symptoms will be quantified using PHQ-2 questionnaire

OTHER OUTCOMES:
New York Heart Association (NYHA) Class | Baseline and 30 days
  Change in NYHA functional class
LV function | Baseline and 30 days
  Echo will be performed to evaluate heart function

IPD SHARING:
Plan to Share IPD: No